CLINICAL TRIAL: NCT05246397
Title: Sugammadex Titration for Reversal of Rocuronium or Vecuronium in Cardiac Surgery Patients
Brief Title: Sugammadex Titration in Cardiac Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, T. Andrew Bowdle, Professor, School of Medicine: Anesthesiology and Pain Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00013925
Record Dates: First submitted 2021-09-23; First posted 2022-02-18 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease; Aorta Disease; Heart Failure
Keywords: neuromuscular blockade; sugammadex; monitoring; rocuronium; vecuronium
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Aortic Diseases; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiac surgery patients (Experimental): Patients undergoing cardiac surgery
  Interventions: Drug: Sugammadex administration

INTERVENTIONS:
Drug: Sugammadex administration — Sugammadex will be given in 50 mg increments every five minutes for reversal of neuromuscular blockade until reaching a train-of-four ratio of 0.9

SUMMARY:
Sugammadex is frequently used to reverse the effects of neuromuscular blocking drugs. The recommended doses are 2 mg/kg or 4 mg/kg depending upon the depth of neuromuscular blockade. Clinical studies and experience have suggested that smaller doses may be effective. The purpose of this observational study is to determine the minimal effective dose of sugammadex by administering 50 mg every 5 minutes until the train-of-four ratio is 0.9 in a cohort of cardiac surgery patients, and to determine the duration of action by measuring the train-of-four every hour for up to 6 hours following reversal.

DETAILED DESCRIPTION:
Neuromuscular blocking drugs are used frequently during general anesthesia. The effects of neuromuscular blocking drugs are measured using a twitch monitor, that stimulates the ulnar nerve and measures the evoked response of the adductor pollicis muscle (thumb flexion), or other intrinsic hand muscle. When a series of 4 twitches is administered, the ratio of the first to the fourth twitch (train-of-four ratio) may be used to gauge the degree of muscle relaxation. A train-of-four ratio of 0.9 or greater is considered to represent adequate recovery from neuromuscular blockade. At the end of surgery, antagonists of neuromuscular blockade are commonly administered to reverse any remaining muscle relaxation. Sugammadex is a highly effective reversal agent of the aminosteroid neuromuscular blockings drugs rocuronium and vecuronium, which are the most commonly used neuromuscular blocking drugs. The recommended dose of sugammadex depends upon the degree of neuromuscular blockade. When at least 1 twitch of the train-of-four is present, the recommended dose of sugammadex is 2 mg/kg. When there are no twitches of the train-of-four present, but at least 1 count of the post tetanic count is present, the recommended dose of sugammadex is 4 mg/kg. However, in several dose ranging studies of sugammadex, and in using sugammadex clinically, we and others have determined that smaller doses of sugammadex, often much less than 2 mg/kg, may be effective producing a train-of-four ratio of 0.9 or greater. Sugammadex binds (encapsulates) aminosteroid neuromuscular blocking drugs tightly and the sugammadex-aminosteroid complex is subsequently cleared by the kidney. Therefore we do not expect that recurrence of neuromuscular blockade would occur, even after small doses of sugammadex, as long as the dose of sugammadex is adequate to produce a train-of-four ratio of 0.9. However, additional studies are needed to confirm that recurrence of neuromuscular blockade does not occur after small doses of sugammadex. The purpose of the proposed study is to test the hypothesis that when sugammadex is titrated in 50 mg increments until the train-of-four ratio is 0.9 or greater, that this train-of-four ratio is maintained and there is no recurrence of neuromuscular blockade.

Neuromuscular blockade will be monitored with EMG (electromyography)-based quantitative twitch monitoring (TwitchView). At the end of cardiac surgery, sugammadex will be administered to reverse neuromuscular blockade, as defined by a train-of-four ratio of 0.9 or greater. The patient will then transported asleep, intubated and ventilated to the intensive care unit where the train-of-four ratio of 0.9 or greater will be confirmed on arrival by the respiratory therapist.

Instead of administering a standard dose of sugammadex 2 mg/kg or 4 mg/kg, sugammadex will be titrated in 50 mg increments every 5 minutes until a train-of-four ratio of 0.9 or greater is reached. Train-of-four ratio will be measured on arrival in the intensive care unit and then hourly for 6 hours or until extubation if extubation occurs in <6 hours. If the train-of-four ratio is less than 0.9 at any time, additional sugammadex will be administered until the train-of-four ratio is 0.9 or greater. The twitch monitoring results in the operating room just prior to reversal, following reversal and hourly in the intensive care unit will be recorded, along with sugammadex doses. The total dose of rocuronium or vecuronium and the time period of neuromuscular blocking drug will also be recorded. Data will either be recorded in real time by study assistants or retrieved from the electronic medical record. The patient's age, gender, and weight will be recorded.

ELIGIBILITY:
Inclusion Criteria

* All cardiac surgery patients

Exclusion Criteria:

* Allergic or other adverse response to sugammadex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T. Andrew Bowdle, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared based on the policy of the journal in which the work is published

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiac Surgery Patients
Started | 100
Completed | 97
Not Completed | 3
Not completed — 3 were excluded due to protocol deviation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (15)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 23
  Male | 73
  Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8
  White | 77
  Other | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 97
Weight [Median (Inter-Quartile Range); unit: kilograms] | 80 [73 to 95]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.9 [0.8 to 1.1]
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 9.2 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Total Dose of Sugammadex Required to Produce a Train-of-four Ratio of >0.9, Categorized as Greater Than or Less Than the Manufacturers Recommended Dose Based on the Train-of-four or Post Tetanic Response Prior to Administration of Sugammadex
Description: Sugammadex will be administered in 50 mg increments every 5 minutes until a train-of-four ratio of at least 0.9 is reached. The total dose of sugammadex for each patient will be categorized as greater than or less than the manufacturers recommended dose
Time Frame: At the completion of surgery and prior to transport to the intensive care unit. The elapsed time from completion of surgery to arrival in the intensive care unit is 30 min to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 97
Participants
  Less than manufacturer's dose | 84
  More than manufacturer's dose | 13

2. Primary Outcome: Duration of Action of Reversal
Description: The train-of-four ratio will be determined upon arrival to the ICU and every hour for 6 hours or until extubation (whichever is less) and categorized as remaining greater than or equal of 0.9, or declining to <0.9 (described as "recurrent" neuromuscular blockade)
Time Frame: On arrival to the intensive care unit and hourly thereafter for 6 hours or until extubation, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 97
Participants
  Recurrent train-of-four ratio <0.9 | 2
  Train-of-four ratio >0.9 | 95

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time that sugammadex administered until the end of twitch monitoring in the intensive care unit, a maximum time of 7 hours.
Arm/Group | Cardiac Surgery Patients
All-Cause Mortality (participants affected / at risk) | 0/97
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05246397/Prot_SAP_000.pdf